CLINICAL TRIAL: NCT04077671
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profiles of CHF6467 After Single and Repeated Ascending Doses in Subjects With Diabetic Neurophatic Foot Ulcers (DFU).
Brief Title: CHF6467 SAD and MAD in Patients With Diabetic Foot Ulcer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: Comac Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLI-06467AA1-01; 2018-001724-19 (EudraCT Number)
Record Dates: First submitted 2019-03-28; First posted 2019-09-04 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Neuropathic Foot Ulcers
Keywords: DFU; Diabetic Foot Ulcers; Diabetic Neuropathic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: SAD - Single Ascending Dose & MAD - Multiple Ascending Dose
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SAD - Cohort A - CHF6467 0.3 µg/mm2 (Experimental): Cohort A: will be administered with CHF6467 0.3 µg/mm2 ulcer area as single dose.
  Interventions: Biological: CHF6467 active
- SAD - Cohort B - CHF6467 1 µg/mm2 (Experimental): Cohort B: will be administered with 1 µg/mm2 ulcer area as single dose.
  Interventions: Biological: CHF6467 active
- SAD - Cohort C - CHF6467 3 µg/mm2 (Experimental): Cohort C: will be administered with 3 µg/mm2 ulcer area as single dose.
  Interventions: Biological: CHF6467 active
- SAD - Cohort D - CHF6467 6 µg/mm2 (Experimental): Cohort D: will be administered with 6 µg/mm2 ulcer area as single dose.
  Interventions: Biological: CHF6467 active
- MAD - Cohort E - CHF6467 0.3 or 1 µg/mm2 (Experimental): Cohort E: will be administered with 0.3 or 1 µg/mm2 ulcer area (total daily dose) as multiple dose (14 days). The dose will be selected based on the SAD results.
  Interventions: Biological: CHF6467 active
- MAD - Cohort F - CHF6467 1 or 3 µg/mm2 (Experimental): Cohort F: will be administered with 1 or 3 µg/mm2 ulcer area (total daily dose) as multiple dose (14 days). The dose will be selected based on the SAD results.
  Interventions: Biological: CHF6467 active

INTERVENTIONS:
Biological: CHF6467 active — CHF6467, is mutated form of the human Nerve Growth Factor (NGF).

SUMMARY:
To assess the safety and tolerability of single and multiple days' topical dosing with CHF6467 in subjects with diabetic foot ulcer (DFU).

DETAILED DESCRIPTION:
This first in human study is designed to investigate the tolerability, safety, pharmacokinetics and preliminarily pharmacodynamics following topical administration of single and multiple ascending doses of CHF6467 in subjects diagnosed with diabetic foot ulcer (DFU).

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure;
2. Male or female subject, aged 18 - 80 years (extremes inclusive), diagnosed with Type I or Type II diabetes mellitus, with glycosylated haemoglobin (HbA1c) ≤ 10%.
3. Female subjects of non-childbearing potential (WONCBP):

   * they must report surgical sterilization (performed at least 6 months prior to screening), or
   * menopause (must have had no regular menstrual bleeding for at least one year prior to screening, age ≥ 45 years and FSH at screening ≥ 40 mIU/ml).
4. Female subject with childbearing potential (WOCBP): they must be using one or more of the following reliable methods of contraception during the study period and at least within 90 days after the last study drug administration:

   1. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
   2. Hormonal contraception (implantable, patch, oral).
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical vaults/caps) with spermicidal foam/gel/film/cream/suppository.
   4. Male Partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
5. Male subjects; they must be using two effective methods of contraception during the entire study period and not donate sperm within 90 days after the last study drug administration.
6. Presence of at least one diabetic foot ulcer meeting the following criteria:

   1. Diagnosed as a full-thickness, neuropathic DFU, located at or distal to the malleolus (excluding ulcers between the toes but including those of the heel)
   2. SAD: Present for 6 weeks to 12 months, and of 3 - 5 cm2 in area following sharp debridement, confirmed at screening.

      MAD: Present for 6 weeks to 12 months, and of 3 - 6 cm2 in area following sharp debridement confirmed at screening, and of 2-5 cm2 after the 2 weeks run-in period with an area reduction compared to screening <50%.
   3. A minimum 1 cm margin between the qualifying study ulcer and any other ulcers on the specified foot.
   4. SAD: Ulcer must have a depth ≥ 5 mm at some point in its area and be graded 1A according to "The University of Texas Staging System for Diabetic Foot Ulcers" (22), with no capsule, tendon or bone exposed and no tunnelling, undermining, or sinus tracts, after the initial sharp debridement, confirmed at screening.

   MAD: Ulcer must have a depth ≥ 5 mm at some point in its area and be graded 1A or 2A according to "The University of Texas Staging System for Diabetic Foot Ulcers" (22), after the initial sharp debridement, confirmed at screening.
7. Subject must be able to hold the target ulcer in such a position and orientation that the study medication can be applied without significant loss of substance through run-off, until the dressing has been applied.
8. Adequate vascular perfusion of the affected limb demonstrated within 30 days prior to screening, as defined by at least one of the following:

   1. Ankle-Brachial Index (ABI) ≥ 0.9 and ≤ 1.2, confirmed by transcutaneous oxygen partial pressure (TcPO2) >50 mmHg
   2. Toe pressure (plethysmography) >50 mmHg
   3. Doppler ultrasound (biphasic or triphasic waveforms) at least on two vessels at the ankle consistent with adequate blood flow to the affected extremity, as determined by SoC.

Exclusion Criteria:

1. For females only: pregnant or lactating female subject, confirmed by a positive serum pregnancy test at screening and a urine test performed on Day -1.
2. Subject with:

   1. Ulcer(s) accompanied by infected cellulitis, osteomyelitis, or clinical signs or symptoms of infection confirmed by a cultural exam made on the material taken off from the ulcer according to the technique described in the guidelines for diagnosis and management of diabetic foot infections of the Infectious Diseases Society of the Americas (IDSA) (19).
   2. Gangrene or necrosis on any part of the affected limb.
   3. Active or chronic Charcot's foot on the study limb.
   4. Planned vascular surgery, angioplasty or thrombolysis or previous revascularization procedure performed within 1 month prior to enrolment.
   5. SD only: Ulcers involving exposure of tendon, bone, or joint capsule (It is acceptable to have ulcers extending through the dermis and into subcutaneous tissue with presence of granulation tissue).
   6. Ulcer(s) of non-diabetic aetiology.
   7. Previous Lisfranc or Chopart's amputations on the same target foot.
   8. Actual or recent (3 weeks) antibiotic therapy for any reason.
   9. Bedridden subjects or subjects with a life expectancy less than one year.
3. Use of any growth factor therapy in the 3 months prior to screening.
4. History of malignancy in the 5 years prior to screening or those with a strong family history of cancer (e.g. familial cancer disorders), with the exception of squamous cell or basal cell carcinoma of the skin that has been definitively treated.
5. Clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, haematological or metabolic disease that is, in the opinion of the Investigator, not stabilised or may otherwise impact subject safety or study results (in cases of doubt, the Sponsor's Clinical Research Physician should be consulted).
6. Subject undergoing haemodialysis or peritoneal dialysis or with chronic renal insufficiency (plasma creatinine > 2 mg/dl).
7. Subject with significantly abnormal key laboratory parameters interfering with the safety of the patient according to the PI judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | SAD: From Day 1 up to Day 28; MAD: From Day 1 up to Day 84;
  During the SAD and the MAD, the number of events and the number and percentage of subjects experiencing TEAEs, treatment emergent ADRs, serious TEAEs, non-serious TEAEs, severe TEAEs, TEAEs leading to discontinuation of study drug and TEAEs leading to death will be presented by treatment.

SECONDARY OUTCOMES:
Pharmacokinetics: AUC0-72h after single administration | SAD: Serial of timepoints until 72 hours post dose
  During the SAD: Dose proportionality of CHF6467 for AUC0-72h, and classical PK parameters will be calculated
Pharmacodynamic: Ulcer area after multiple administration | MAD: From Day 1 to Days 4, 7, 10, 14, 17, 21, 24, 28, 31, 35, 38, 42, 45, 49, 52, 56, 59, 63, 66, 70, 73, 77, 80 and 84
  MAD: Ulcer area measurements expressend in cm2 over time after multiple administration
Pharmacokinetics: AUC0 to infinit after multiple administration | MAD: Serial of timepoints at Day 1, Day 2, Day 4, Day 7, Day 10, Day 13, Day 14, Day 21 and Day 28
  During the MAD: Dose proportionality of CHF6467 for AUC 0 to infinit, and classical PK parameters will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Iliya Lozev, MD, Principal Investigator — Comac Medical
Locations (1):
- Comac Medical Ltd., Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2018-001724-19/results
- See also: Lay Summaries of study results available in the CHIESI Clinical Study Register — https://www.chiesi.com/en/chiesi-clinical-study-register/